CLINICAL TRIAL: NCT06921135
Title: The Impact of Nutritional Intervention in Young Children in PPR Lembah Subang 1: A Retrospective Study
Brief Title: Nutrition of Urban-poor Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Version 1.0
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Dietary Assessment; Growth; Nutritional Assessment
Keywords: Dietary diversity; Food supplement; malnutrition in children; Healthy food choice; sugar sweetened beverages and food
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Dietary Supplements; Food

STUDY DESIGN:
Intervention Model Description: The study will be a retrospective pre-post interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community (Active Comparator): Regular food supplementation.
  Interventions: Dietary Supplement: supplementation, food
- Child Health Clinic (No Intervention): No food supplementation.

INTERVENTIONS:
Dietary Supplement: supplementation, food — Supplementation of fresh foods
  Arms: Community

SUMMARY:
The investigators undertook a program to promote the consumption of healthy foods and reduce the prevalence of malnutrition of children below the age of 5 years in an urban-poor community, by 10% year-on-year through nutrition education and the provision of healthy food. The main purpose of the study is to determine the impact of these nutrition intervention programs on the nutritional status of children under-5 in Selangor.

This retrospective pre-post intervention study will use data collected from 2 previous studies that were carried out between July 2020 to May 2021 (Eat Healthy Project 1.0) and March 2022 to December 2023 (Eat Healthy Project 2.0). The 2 studies had been approved by the Medical Research and Ethics Committees of University Malaya Medical Centre (UMMC) and the Ministry of Health, Malaysia and registered with the National Medical Research Registry (NMRR).

The main outcome measures were:

1. Improved dietary practices, in particular, an increase in the proportion of children who meet the minimum dietary diversity score of 5 food groups, post-intervention.
2. An increase in proportion of children consuming fruits and vegetables and a decrease in proportion of children consuming sugar-sweetened foods and beverages post-intervention.
3. A decrease in prevalence of malnutrition - underweight, wasting and stunting. The comparator will be urban-poor children attending a Child Health clinic who had received nutritional education but no provision of food supplementation.

DETAILED DESCRIPTION:
The primary objectives:

1. To compare dietary diversity practices of children, based on the WHO 8 food groups and 24-hour dietary recall, pre- and post-intervention.
2. To compare consumption of fresh foods, sugar-sweetened foods and beverages pre- and post-intervention.

   The secondary objectives:
3. To compare the weight-for-age z-scores of children pre- and post-intervention.
4. To compare the height-for-age z-scores of children pre- and post-intervention.
5. To compare the prevalence of malnutrition: underweight, stunting and wasting pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* children aged under 5 years enrolled at PPR Lembah Subang 1 or
* children aged under 5 years enrolled at the Child Health Clinic, Universiti Malaya Medical Center

Exclusion Criteria:

* Children with low birth weight (<2.5 kg)
* Children born pre-term (<37 weeks gestation) and
* Children with chronic illnesses or severe malnutrition.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2020-07-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Minimum Dietary diversity score | Pre and post intervention, at least 4 months interval
  The percentage of children who achieved the minimum dietary diversity score of 5 food groups, based on WHO 8 food groups and 24-hour dietary recall.
Consumption of healthy foods | Pre and post intervention, at least 4 months interval
  The percentage of children who consume fresh fruits and/or vegetables pre- and post-intervention.
Consumption of unhealthy foods | Pre and post intervention, at least 4 months interval
  The percentage of children who consume sugar-sweetened foods or beverages.

SECONDARY OUTCOMES:
Child's weight z-scores | Pre and post intervention, at least 4 months interval
  Weight is measured in kilograms Weight will be adjusted for age and sex, i.e., Weight for age Z-score
Child's Height z-scores | Pre and post intervention, at least 4 months interval
  Height is measured centimeters, adjusted for age and sex: Height-for-age Z-score

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti of Malaya Medical Center, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
IPD used in results publication
Supporting Information: Study Protocol, ICF
Time Frame: December 2025 to November 2026
Access Criteria: To request for access from the PI
URL: https://data.mendeley.com/research-data/?

REFERENCES:
- See also: The Role of Nutrition in Brain Development: The Golden Opportunity of the "First 1000 Days" — https://doi.org/10.1016/j.jpeds.2016.05.013
- See also: Advocacy for Improving Nutrition in the First 1000 Days to Support Childhood Development and Adult Health — https://pubmed.ncbi.nlm.nih.gov/29358479/
- See also: Moursi, M., Arimond, M., Dewey, K., Trèche, S., Ruel, M., & Delpeuch, F. (2008). Dietary Diversity Is a Good Predictor of the Micronutrient Density of the Diet of 6- to 23-Month-Old Children in Madagascar. — https://doi.org/10.3945/jn.108.093971
- See also: World Health Organization. Indicators for assessing infant and young child feeding practices Part 1: Definitions. Geneva: WHO; 2008. — https://apps.who.int/iris/bitstream/handle/10665/43895/9789241596664_eng.pdf;sequence=1